CLINICAL TRIAL: NCT02871050
Title: The Castleman Disease Collaborative Network Biobank: A Collection of Biospecimens and Clinical Data to Facilitate Research
Brief Title: Castleman Disease Collaborative Network Biobank
Acronym: "Castlebank"
Status: Withdrawn | Type: Observational
Why Stopped: An alternative Biobank Project was initiated.
Sponsor: Castleman Disease Collaborative Network (Other)
Responsible Party: Sponsor
Other Study IDs: #31132/1
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Castleman Disease; Castleman's Disease; Giant Lymph Node Hyperplasia; Angiofollicular Lymph Hyperplasia; Angiofollicular Lymph Node Hyperplasia; Angiofollicular Lymphoid Hyperplasia; GLNH; Hyperplasia; Giant Lymph Node
Keywords: Biobank; biorepository; Castlebank; Castleman Disease; CD; MCD; iMCD; Castleman; Castleman's Disease; multicentric Castleman's disease; multicentric Castleman disease; Angiofollicular Lymph Hyperplasia
MeSH Terms: conditions — Castleman Disease; Hyperplasia; Macular dystrophy, corneal type 1; Multi-centric Castleman's Disease | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Lymph node and/or bone marrow slides and/or tissue blocks, saliva, whole blood, and serum will be collected both prospectively and retrospectively.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Castleman Disease Patients: Potential study participants may be of any age, gender, or ethnicity who have been diagnosed with Castleman disease.
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — Excess blood sample tubes and/or buccal swabs or saliva will have DNA and RNA extracted and serum and plasma separated out to be stored for future research purposes based on the results of this preliminary research.

SUMMARY:
The purpose of this study is to create a biobank, which collects, stores, and distributes samples of human tissues, blood, and related health information to qualified scientists, in order to help doctors and researchers better understand why Castleman Disease occurs and develop ways to better treat and prevent it.

DETAILED DESCRIPTION:
The CDCN proposes to establish a biobank and associated clinical data for Castleman disease. Tissue and fluid (blood and saliva) samples will be collected both prospectively and retrospectively. Blood or saliva samples may also be collected from relatives of Castleman patients. Because of the scarcity of these samples, it will be necessary to make efforts to access all available cases. Many cases will occur at hospitals that do not have an existing relationship with the CDCN and may not have experience with tissue procurement; however, this is the only way to obtain the vast majority of samples. Samples may be used immediately, banked for future use, or further processed into DNA, cell lines, tissue microarrays, etc.

The samples will be stored at Precision for Medicine, a biorepository company that specializes in collection, processing, storage and distribution of biospecimens. Only researchers (US or international) who have applied to the CDCN and have been approved by the Biobank Advisory Board will be eligible to access biospecimens and/or data. The Biobank Advisory Board will be comprised of clinicians and scientists with experience in clinical and investigational practices in Castleman Disease.

ELIGIBILITY:
Inclusion Criteria

* Potential study participants may be of any age, gender, or ethnicity who have been diagnosed with Castleman disease

Exclusion Criteria

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Castleman Disease patients worldwide
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Samples Collected | 3 years
  Number of samples collected across different subgroups (e.g. blood products, lymph node)

CONTACTS AND LOCATIONS:
Overall Officials: David C Fajgenbaum, MD, MBA, MSc, Principal Investigator — Executive Director of Castleman Disease Collaborative Network
Locations (1):
- Castleman Disease Collaborative Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified Researchers, who apply for access to the database and are subsequently approved, will be given access to a limited dataset with direct identifiers removed in an Excel compatible file format or single SAS data files. The Biobank Advisory Board will review applications from qualified researchers on an ongoing basis.

REFERENCES:
- [Background] Liu AY, Nabel CS, Finkelman BS, Ruth JR, Kurzrock R, van Rhee F, Krymskaya VP, Kelleher D, Rubenstein AH, Fajgenbaum DC. Idiopathic multicentric Castleman's disease: a systematic literature review. Lancet Haematol. 2016 Apr;3(4):e163-75. doi: 10.1016/S2352-3026(16)00006-5. Epub 2016 Mar 17. PMID 27063975
- [Background] Fajgenbaum DC, van Rhee F, Nabel CS. HHV-8-negative, idiopathic multicentric Castleman disease: novel insights into biology, pathogenesis, and therapy. Blood. 2014 May 8;123(19):2924-33. doi: 10.1182/blood-2013-12-545087. Epub 2014 Mar 12. PMID 24622327
- See also: website includes information on Castleman Disease — http://www.cdcn.org
- See also: Please visit this link to sign-up and contribute samples! — http://www.cdcn.org/samples